CLINICAL TRIAL: NCT07402564
Title: The Effect of Mindfulness-based Psychoeducation Program on Job Stress, Job Satisfaction and Job Performance Among Nurses: A Randomized Controlled Study
Brief Title: Mindfulness-Based Program for Nurses' Stress, Satisfaction, and Performance
Acronym: MIND-NURSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kamuran Cerit (Other)
Responsible Party: Sponsor-Investigator, Kamuran Cerit, Assistant Professor, PhD, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDU-KC-MINDFULNESS
Record Dates: First submitted 2025-11-19; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Job Stress; Job Satisfaction; Work Performance
Keywords: Mindfulness; mindfulness-based intervention; job stress; job satisfaction; job performance; nurses; randomized controlled trial
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group, which will receive the mindfulness-based psychoeducation program, or the control group, which will receive no intervention during the study period. Both groups will be assessed at baseline, post-intervention, and at 3-month follow-up.
Who Masked: Outcomes Assessor
Masking Description: Randomization, intervention delivery, and outcome assessment will be conducted by three different researchers to maintain role separation. The researcher responsible for randomization will generate and assign the allocation sequence but will not be involved in intervention delivery or data assessment. The researcher delivering the mindfulness-based intervention will know group assignments but will not participate in data collection or analysis. The outcomes assessor, who is responsible for data collection and statistical analysis, will remain blinded to group assignments throughout the study and will not have access to the randomization list or any information that could reveal participant allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Psychoeducation Program (Experimental): The intervention group will consist of nurses assigned to three separate groups, each including 10-12 participants. The mindfulness training program will be delivered once per week for 90 minutes, for a total of four sessions. To prevent information sharing with the control group, participants will provide informed consent agreeing not to discuss the training content during the study period. Assessments will be administered at Week 4 (immediately after the final session) and at Week 16 (12 weeks after the final session).
  Interventions: Behavioral: Mindfulness-Based Psychoeducation Program
- Control Group (No Intervention): Participants in the control group (Wait-List Control) will not receive the intervention during the study period but will complete all assessments at Week 0 (Baseline), Week 4, and Week 16. After all data collection is completed, they will be offered the mindfulness program.This design ensures that all participants have access to the program while maintaining a proper control comparison.

INTERVENTIONS:
Behavioral: Mindfulness-Based Psychoeducation Program — The mindfulness-based psychoeducation program, developed by an Associate Professor in psychiatric nursing, consists of four weekly 90-minute sessions tailored to nurses' working conditions. It includes selected exercises from Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy programs, along with homework to practice skills between sessions. The program's content and objectives were validated by ten mindfulness experts using the Lawshe method and Content Validity Ratios.
  Arms: Mindfulness-Based Psychoeducation Program

SUMMARY:
Nurses often work in busy and stressful hospital environments, which can affect their well-being, job satisfaction, and work performance. Mindfulness is a set of practices that help individuals focus on the present moment and cope better with stress. Mindfulness-based programs have been shown to reduce stress and improve emotional well-being in healthcare workers, but their effects on nurses' job satisfaction and work performance are not yet well understood.

This study aims to examine whether a mindfulness-based psychoeducation program can reduce job stress and improve job satisfaction and job performance among nurses. The study will include nurses working in a public hospital in Isparta, Turkey. Participants will be randomly assigned to either an intervention group that receives the mindfulness program or a control group. All participants will complete assessments before the program, after the program, and again three months later.

The findings of this study are expected to provide useful information on whether mindfulness training can improve nurse's important work-related outcomes.

DETAILED DESCRIPTION:
Mindfulness has long been an important area of research in clinical psychology, and its use has expanded into organizational settings as evidence grows regarding its positive effects on employees' well-being and work-related outcomes. Nurses, who often work under heavy workload, emotional demands, and stressful conditions in hospital environments, are among the occupational groups that may benefit most from such interventions. High levels of work stress among nurses can negatively influence their psychological, physiological, and social well-being, and can reduce job satisfaction and work performance.

Although previous studies have examined the impact of mindfulness-based programs on outcomes such as stress, burnout, empathy, depressive symptoms, and quality of work life among nurses, the evidence regarding their effects on job satisfaction is limited and inconsistent. Moreover, mindfulness-based interventions have rarely been evaluated in relation to the multidimensional nature of nurses' job performance. There remains a need for well-designed studies that examine how mindfulness training may influence nurses' job-related outcomes more comprehensively.

This study aims to address this gap by evaluating the effects of a mindfulness-based psychoeducation program on job stress, job satisfaction, and job performance among nurses working in a major public hospital in Isparta, Turkey. The study will employ a randomized controlled design with baseline, post-intervention, and three-month follow-up assessments. Nurses will be randomly allocated to an intervention group, which will participate in the mindfulness-based psychoeducation program, or to a control group that will not receive any intervention during the study period.

The intervention includes structured psychoeducational content and mindfulness practices tailored for healthcare professionals, focusing on developing present-moment awareness, improving coping skills, and enhancing emotional balance in demanding clinical environments. By assessing changes across multiple time points, the study aims to provide a more complete understanding of the program's short-term and sustained effects.

The findings are expected to contribute to the literature by offering clearer evidence on whether mindfulness-based programs can improve nurses' job stress and key job-related outcomes, particularly job satisfaction and multidimensional job performance, which have been insufficiently explored in previous research.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as a staff nurse in the hospital's clinical units.
* Willing to voluntarily participate in the study.

Exclusion Criteria:

* Previous participation in any mindfulness-based program.
* Presence of a major psychiatric disorder or currently receiving psychiatric medication or psychotherapy.
* Active medical condition that prevents participation in the program (e.g., malignancy).
* Currently experiencing bereavement.
* Holding managerial or head nurse positions, due to different roles and responsibilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Job stress | Baseline, Week 4, Week 16
  Job stress will be measured using the General Work Stress Scale (GİSÖ), adapted into Turkish by Teleş (2021). The scale consists of 9 items rated on a 5-point Likert scale (1 = Never, 5 = Always) and evaluates general work-related stress among nurses.
Job Satisfaction | Baseline, Week 4, Week 16
  Job satisfaction will be assessed using the Short Form Minnesota Satisfaction Questionnaire (SFMSQ), Turkish version by Baycan (1985). The scale includes 20 items rated on a 5-point Likert scale (1 = Very dissatisfied, 5 = Very satisfied) and measures overall job satisfaction, intrinsic satisfaction, and extrinsic satisfaction.
Individual Job Performance | Baseline, Week 4, Week 16
  Individual job performance will be measured using the Individual Job Performance Scale, Turkish adaptation (Köroğlu Kaba & Öztürk, 2021). The 14-item scale assesses three domains: task performance (items 1-5), contextual performance (items 6-11), and counterproductive work behavior (items 12-14), rated on a 5-point Likert scale (1 = Rarely, 5 = Always).

SECONDARY OUTCOMES:
Mindfulness Level | Baseline, Week 4, Week 16
  Mindfulness will be measured using the Mindful Attention Awareness Scale (MAAS) (Brown & Ryan, 2003). The scale contains 15 items and provides a single total score reflecting the general tendency to be attentive and aware of present-moment experiences in daily life.
Demographic Information | Baseline
  Demographic characteristics including age, gender, education, marital status, work experience, and department will be collected using a researcher-developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kamuran Cerit, Principal Investigator — Süleyman Demirel University, Faculty of Health Sciences, Department of Nursing

IPD SHARING:
Plan to Share IPD: Undecided
Any potential future sharing would follow strict anonymization and ethical approval procedures to protect participant confidentiality.

REFERENCES:
- [Background] Hilcove K, Marceau C, Thekdi P, Larkey L, Brewer MA, Jones K. Holistic Nursing in Practice: Mindfulness-Based Yoga as an Intervention to Manage Stress and Burnout. J Holist Nurs. 2021 Mar;39(1):29-42. doi: 10.1177/0898010120921587. Epub 2020 May 27. PMID 32460584
- [Background] Parvaresh, M., Taghinezhad, N., Amirfakhraei, A., & Sabahizadeh, M. (2023). Effectiveness of Mindfulness-Based Cognitive Flexibility Training on Nurses' Job Satisfaction. Journal of Assessment and Research in Applied Counseling, 5(2), 146-155.
- [Background] Ghawadra, S.F., Abdullah, K.L., Choo, W.Y., Danaee, M., & Phang, C.K. (2020). The effect of mindfulness-based training on stress, anxiety, depression, and job satisfaction among ward nurses: A randomized control trial. Journal of Nursing Management, 28(5), 1088-1097.
- [Background] Çalışkan, B.B., Güneş, A., Tekin, Y.E., Ayvaz, M.Y., & Kızıl, H. (2024). The effect of conscious mindfulness-based program (MBP) applied to emergency nurses on their anxiety and quality of life: A randomized controlled study. Journal of Psychiatric Nursing, 15(3), 225-233.
- [Background] Bazarko, D., Cate, R.A., Azocar, F., Kreitzer, M.J. (2013). The impact of an innovative mindfulness-based stress reduction program on the health and well-being of nurses employed in a corporate setting. J Workplace Behav Health, 28(2),107-33.
- [Background] Alfurjani AM, Al-Hammouri MM, Rababah JA, Alhawatmeh HN, Hall LA. The effect of a mindfulness-based intervention on stress overload, depression, and mindfulness among nurses: A randomized controlled trial. Worldviews Evid Based Nurs. 2024 Feb;21(1):34-44. doi: 10.1111/wvn.12695. Epub 2023 Dec 11. PMID 38083806